CLINICAL TRIAL: NCT05174975
Title: Tri-Service General Hospital, Department of Internal Medicine
Brief Title: Effectiveness of App-based Positive Psychological Intervention on Patients Newly Diagnosed With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Chieh-Hua Lu, director, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B202105141
Record Dates: First submitted 2021-11-16; First posted 2022-01-03 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; self-care behaviors; quality of lofe
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-based Positive Psychological Intervention group (Experimental): The intervention will be conducted on the app, including 2-week PPI, diabetes-related health education, physical records, and online consultation.
  Interventions: Behavioral: App-based Positive Psychological Intervention
- control group (No Intervention): usual care which will educated by certificated educators in terms of self-management

INTERVENTIONS:
Behavioral: App-based Positive Psychological Intervention — The PPI has included a 12-week PPI lessons. Each lesson has separated into 3 parts: introduction, activity, and feedback. Diabetes-related health education will include the basic knowledge of diabetes, diet, and exercise related videos. Physical records include record of daily blood sugar, blood pressure, HbA1c, diet, and exercise. In terms of dietary records, the amount of carbohydrates of each food will be calculate automatically after documented. Exercise records documents the burn of calories of each exercise (per 30 minutes). Both unit of dietary and exercise are based on Health Promotion Administration's criteria in Taiwan. Moreover, participants are available to have one-on-one instant online consultation with their diabetes educators via App.
  Arms: App-based Positive Psychological Intervention group

SUMMARY:
The aim of this experimental study is to explore the effectiveness of app-based positive psychology intervention (PPI) on patients newly diagnosed with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Positive psychological constructs (PPCs), such as optimism, gratitude, self-efficacy, and resilience have been considered to positively impact adherence and self-care behaviour of patients with type 2 diabetes (T2DM). Moreover, diabetes self-care behaviours would be consistently improved as the PPCs have strengthened. Based on systematic reviews, the positive psychological intervention has significantly improved positive emotions, quality of life, self-efficacy, depression, optimism, gratitude, and well-being of patients with T2DM The strengthen of PPCs could be regarded as a strategy for improving type 2 diabetes self-management.

Positive psychology intervention (PPI) emphasis enhancing PPCs via consciousness raising and enhancing personal strengths. With the systemic practice of PPI, it develops individual positive cognition and emotions. A previous Internet-based intervention study found that people have been taught positive emotional skills shown a significantly lower depression level than those having the daily emotional diary. Additionally, a one-group pre-post test study found that both optimism and gratitude have significantly increased after a 12-week phone-based PPI in patients with T2DM. Another one-group pretest-posttest study demonstrated that optimism and well-being had significantly increased after a 12-week PPI. Furthermore, optimism, gratitude, frustrated, depressive, and distress, diabetes self-care and health behaviours adherence have obvious improved. A recent study demonstrated that self-care behaviour and diet behaviour had significantly improved after a 16-week phone-based psychological-motivational interviewing intervention among the patients with Type 2 diabetes (T2DM) with 8 years duration of diabetes. Although previous studies have demonstrated the effectiveness of PPI on PPCs, only few studies investigate the impact on patients newly diagnosed with T2DM. Thus, the aim of this study is to explore the effectiveness of app-based PPI on patients newly diagnosed with T2DM.

Patients newly diagnosed with T2DM of an endocrinology clinic in a medical center in northern Taiwan are assigned to the experimental group (n=57), while patients at an endocrinology clinic in southern Taiwan are assigned to the control group (n=113). Experimental group will have a 3-month App-based intervention, while the control group only have a diabetes-related health education by certificated diabetes educators. Outcome variables will be collected from medical records and self-reported questionnaires. A Generalized Estimation Equation (GEE) is used to compare the changing amount of outcome variables from baseline to week at the end of intervention, to 3 months, and to 9 months post-intervention between a control group and experimental group. A p-value <.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with T2DM less than 6 months
* aged 20 to 64
* controlling diabetes through oral medication or insulin injection
* able to use Android phone

Exclusion Criteria:

* unable to communicate with language or having mental illness

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life | At baseline and 1 week, 3 months and 9 months after the interventiont
  A 15-item Quality of Life Scale will be used to measure quality of life. Each item is rated from 0 (Never) to 4(Always), with higher scores indicating a higher quality of life.
Change in Self-care behaviour | At baseline and 1 week, 3 months and 9 months after the intervention
  A 17-item Diabetes Self-care Behaviour Scale-Chinese version will be used to measure. Each item is rates from 0 (never) to 4 (always). The higher score indicates a greater execution in self-care behaviours.
Change in Glycosylated hemoglobin(HbA1c) levels | At baseline and 1 week, 3 months and 9 months after the intervention
  Collect from medical records

SECONDARY OUTCOMES:
Change in Diabetes Distress | At baseline and 1 week, 3 months and 9 months after the intervention
  A 8-item short form of Problem Areas in Diabetes scale in Chinese version will be used to measure. Each items is rated from 0 (not a problem) to 4 (very serious problem). The higher score indicates a greater level of diabetes distress.
Change in Optimism | At baseline and 1 week, 3 months and 9 months after the intervention
  A 6-item Life Orientation Test-Revised will be used to measure. Each item is rated from 0 as strongly disagree to 4 as strongly agree. The higher scores indicates higher dispositional level of optimism.
Change in Gratitude | At baseline and 1 week, 3 months and 9 months after the intervention
  A 6-item Gratitude Questionnaire will be used to measure. Each item is rated from 1 (strongly disagree) to 7 (strongly agree). The higher score indicates higher gratitude disposition.
Change in Diabetes Self-efficacy | At baseline and 1 week, 3 months and 9 months after the interventiont
  A 14-item Diabetes Self-efficacy scale will be used to measure. Each item is rated from 0 as "Extremely unconfident" to 4 as "80% to 100% confident". The higher score indicates the better self-efficacy.
Change in Diabetic Positive Characteristics | At baseline and 1 week, 3 months and 9 months after the intervention
  A 20-item Diabetic Positive Characteristic Scale will be used to measure. Each item is rated from 1 as "strongly disagree" to 5 as "strongly agree". The overall score is 100 points, with higher scores indicating greater likelihood of positive characteristics disposition.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Hua Lu, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
depend on the finding and process of publication

REFERENCES:
- [Background] Celano CM, Beale EE, Moore SV, Wexler DJ, Huffman JC. Positive psychological characteristics in diabetes: a review. Curr Diab Rep. 2013 Dec;13(6):917-29. doi: 10.1007/s11892-013-0430-8. PMID 24048687
- [Background] Celano CM, Gianangelo TA, Millstein RA, Chung WJ, Wexler DJ, Park ER, Huffman JC. A positive psychology-motivational interviewing intervention for patients with type 2 diabetes: Proof-of-concept trial. Int J Psychiatry Med. 2019 Mar;54(2):97-114. doi: 10.1177/0091217418791448. Epub 2018 Aug 16. PMID 30114958
- [Background] Cohn MA, Pietrucha ME, Saslow LR, Hult JR, Moskowitz JT. An online positive affect skills intervention reduces depression in adults with type 2 diabetes. J Posit Psychol. 2014 Jan 1;9(6):523-534. doi: 10.1080/17439760.2014.920410. PMID 25214877
- [Background] Dubois CM, Beach SR, Kashdan TB, Nyer MB, Park ER, Celano CM, Huffman JC. Positive psychological attributes and cardiac outcomes: associations, mechanisms, and interventions. Psychosomatics. 2012 Jul-Aug;53(4):303-18. doi: 10.1016/j.psym.2012.04.004. PMID 22748749
- [Background] Hsu HC, Lee YJ, Wang RH. Influencing Pathways to Quality of Life and HbA1c in Patients With Diabetes: A Longitudinal Study That Inform Evidence-Based Practice. Worldviews Evid Based Nurs. 2018 Apr;15(2):104-112. doi: 10.1111/wvn.12275. Epub 2018 Feb 14. PMID 29443437
- [Background] Hsu HC, Chang YH, Lee PJ, Chen SY, Hsieh CH, Lee YJ, Wang RH. Developing and psychometric testing of a short-form problem areas in diabetes scale in chinese patients. J Nurs Res. 2013 Sep;21(3):212-8. doi: 10.1097/01.jnr.0000432048.31921.e2. PMID 23958611
- [Background] Huffman JC, DuBois CM, Millstein RA, Celano CM, Wexler D. Positive Psychological Interventions for Patients with Type 2 Diabetes: Rationale, Theoretical Model, and Intervention Development. J Diabetes Res. 2015;2015:428349. doi: 10.1155/2015/428349. Epub 2015 Apr 29. PMID 26064980
- [Background] Huffman JC, Feig EH, Millstein RA, Freedman M, Healy BC, Chung WJ, Amonoo HL, Malloy L, Slawsby E, Januzzi JL, Celano CM. Usefulness of a Positive Psychology-Motivational Interviewing Intervention to Promote Positive Affect and Physical Activity After an Acute Coronary Syndrome. Am J Cardiol. 2019 Jun 15;123(12):1906-1914. doi: 10.1016/j.amjcard.2019.03.023. Epub 2019 Mar 19. PMID 30979409
- [Background] Lee YJ, Shin SJ, Wang RH, Lin KD, Lee YL, Wang YH. Pathways of empowerment perceptions, health literacy, self-efficacy, and self-care behaviors to glycemic control in patients with type 2 diabetes mellitus. Patient Educ Couns. 2016 Feb;99(2):287-94. doi: 10.1016/j.pec.2015.08.021. Epub 2015 Sep 2. PMID 26341940
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629
- [Background] Miller CK, Kristeller JL, Headings A, Nagaraja H. Comparison of a mindful eating intervention to a diabetes self-management intervention among adults with type 2 diabetes: a randomized controlled trial. Health Educ Behav. 2014 Apr;41(2):145-54. doi: 10.1177/1090198113493092. Epub 2013 Jul 12. PMID 23855018
- [Background] Moskowitz JT, Carrico AW, Duncan LG, Cohn MA, Cheung EO, Batchelder A, Martinez L, Segawa E, Acree M, Folkman S. Randomized controlled trial of a positive affect intervention for people newly diagnosed with HIV. J Consult Clin Psychol. 2017 May;85(5):409-423. doi: 10.1037/ccp0000188. Epub 2017 Mar 23. PMID 28333512
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Steinhardt MA, Brown SA, Dubois SK, Harrison L Jr, Lehrer HM, Jaggars SS. A resilience intervention in African-American adults with type 2 diabetes. Am J Health Behav. 2015 Jul;39(4):507-18. doi: 10.5993/AJHB.39.4.7. PMID 26018099

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT05174975/Prot_SAP_000.pdf